CLINICAL TRIAL: NCT01103973
Title: The Impact of Distress on the IVF Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070076
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Infertility
Keywords: IVF, Mind/Body
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Spa Certificate) (Placebo Comparator): For every three months in the study control subjects received $50 spa gift certificates.
  Interventions: Behavioral: Control
- Mind/Body Program (Experimental): Ten week group mind/body program. Skills include relaxation training, cognitive strategies, and lifestyle modifications.
  Interventions: Behavioral: Mind/Body Program

INTERVENTIONS:
Behavioral: Mind/Body Program — Ten week group mind/body program
  Arms: Mind/Body Program
Behavioral: Control — Spa gift certificates
  Arms: Control (Spa Certificate)

SUMMARY:
Stress is a primary reason why in vitro fertilization (IVF) patients drop out of treatment, and it may have a detrimental impact on pregnancy rates, yet there is minimal published research on the efficacy of structured skills-based psychological interventions with assisted reproductive technology (ART) patients. The objective of this study is to determine if women who are randomized to a mind/body (MB) program prior to starting their first IVF cycle will have higher pregnancy rates than controls (C).

This is a randomized, controlled prospective study conducted at a private academically-affiliated infertility clinic and includes 143 women ages 40 and below scheduled to undergo their first IVF cycle. Subjects are randomized via computer generated random numbers table to a 10 session mind/body program or a control group and followed for two IVF cycles. The primary outcome measure is clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Female Boston IVF infertility patient
* Age 21-40 years
* Day 3 FSH level 12 mIU/ml or below
* Day 3 E2 level 80 pg/ml or below
* Using own eggs (not an egg donor)
* Daily access to the internet
* Able to read, understand, and sign the informed consent in English

Exclusion Criteria:

* Prescription antipsychotic medication
* Diagnosis of borderline or narcissistic personality disorder
* Previous participation in a MB group

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice D Domar, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domar AD, Rooney KL, Wiegand B, Orav EJ, Alper MM, Berger BM, Nikolovski J. Impact of a group mind/body intervention on pregnancy rates in IVF patients. Fertil Steril. 2011 Jun;95(7):2269-73. doi: 10.1016/j.fertnstert.2011.03.046. Epub 2011 Apr 15. PMID 21496800

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 women withdrew or were ineligible for the study. The reasons for withdrawal were: 1) no longer eligible owing to no subsequent IVF cycle (15 patients); 2) too great a time commitment (15 patients); 3) noncompliance with study requirements (7 patients); 4) dislike of study tasks (6 patients); and 5) other (3 patients).
Period: Overall Study
Arm/Group | Control (Spa Certificate) | Mind/Body Program
Started | 51 | 46
Completed | 51 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Spa Certificate) | Mind/Body Program | Total
Number analyzed (Participants) | 51 | 46 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (3.8) | 34 (3.7) | 34 (3.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 46 | 97
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rates
Description: Presence of normal fetal heart rate and fetal size at 7 weeks gestation.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Control (Spa Certificate) | Mind/Body Program
Number analyzed (Participants) | 51 | 46
percentage of participants | 20 | 52

2. Secondary Outcome: Pregnancy Rate Based on Psychological Status Assessed by the Beck Depression Inventory (BDI)
Description: Psychological status is assessed by the Beck Depression Inventory (BDI). The scores range from 0 to 63; a score of 0 being no depression and 63 being severely depressed. Our cut-off for normal was a score of 12 or less, and those with a score of 13 or greater were considered to have symptoms of depression.
Time Frame: 1 year
Population: Subjects were evaluated before IVF cycle 1 and cycle 2 if applicable. The N varies per cycle as some patients withdrew from the study or did not have a second cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Spa Certificate) | Mind/Body Program
Number analyzed (Participants) | 51 | 46
Participants
  Pregnancy Rate for BDI ≥ 12 at Cycle 1: number analyzed (Participants) | 33 | 33
  Pregnancy Rate for BDI ≥ 12 at Cycle 1 | 15 | 12
  Pregnancy Rate for BDI ≤ 12 at Cycle 2: number analyzed (Participants) | 14 | 18
  Pregnancy Rate for BDI ≤ 12 at Cycle 2 | 4 | 9
  Pregnancy Rate for BDI ≥ 13 at Cycle 1: number analyzed (Participants) | 18 | 13
  Pregnancy Rate for BDI ≥ 13 at Cycle 1 | 7 | 8
  Pregnancy Rate for BDI ≥ 13 at Cycle 2: number analyzed (Participants) | 6 | 3
  Pregnancy Rate for BDI ≥ 13 at Cycle 2 | 0 | 2

ADVERSE EVENTS:
Arm/Group | Control (Spa Certificate) | Mind/Body Program
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/46
Other Adverse Events (participants affected / at risk) | 0/51 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No